CLINICAL TRIAL: NCT01926184
Title: Randomized Controlled Trial of an Integrative Intervention for Non-Treatment-Seeking Meth Users
Brief Title: RCT of an Integrative Intervention for Non-Treatment-Seeking Meth Users
Acronym: ARTEMIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01DA033854 (NIH); R01DA033854 (NIH)
Record Dates: First submitted 2013-08-16; First posted 2013-08-20 (Estimated); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: HIV/AIDS; Stimulant Use Disorders
Keywords: HIV/AIDS; Treatment as Prevention; Methamphetamine; Cocaine; HIV viral Load
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ARTEMIS+CM (Experimental): This is a 5-session, individually delivered intervention that is designed to enhance positive affect. It is designed to boost and extend the effectiveness of contingency management (CM).
  Interventions: Behavioral: Affect Regulation Treatment to Enhance Meth Intervention Success (ARTEMIS); Behavioral: Contingency Management (CM)
- Attention-Control+CM (Placebo Comparator): Attention-matched, 5-session control condition consisting of brief-self report psychological measures and neutral writing exercises. Contingency management (CM) is also administered to this arm.
  Interventions: Behavioral: Contingency Management (CM)

INTERVENTIONS:
Behavioral: Affect Regulation Treatment to Enhance Meth Intervention Success (ARTEMIS) — 5-session integrative intervention to improve positive affect as well as boost and extend the effectiveness of contingency management (CM).
  Arms: ARTEMIS+CM
Behavioral: Contingency Management (CM) — 12-week CM protocol that provides escalating monetary reinforcement for biological evidence of methamphetamine abstinence. Delivered as the standard of care for non-treatment-seeking methamphetamine-using MSM in San Francisco. Delivered to both the intervention and attention-control arms
  Other Names: Positive Reinforcement Opportunity Project (PROP)

SUMMARY:
In the era of HIV treatment as prevention (TasP), efforts are needed to identify evidence-based combination prevention approaches that achieve greater decreases HIV viral load among populations that are more likely to engage in HIV transmission risk behavior. Because methamphetamine-using men who have sex with men (MSM) are at greater risk for acquiring and transmitting HIV, interventions targeting stimulant use in this population of high-risk men could boost the effectiveness of TasP. At present, only conditional cash transfer approaches such as contingency management (CM) have demonstrated short- term efficacy in reducing stimulant use among substance-using MSM who are not actively seeking formal treatment. The proposed RCT will examine the efficacy of a positive affect intervention that is designed to optimize the effectiveness of CM to achieve long-term reductions in stimulant use and HIV viral load in this population. the team will examine the efficacy of this integrative intervention in a randomized controlled trial (RCT) with 110 HIV-positive, methamphetamine-using MSM. After enrolling in CM, participants will be randomized to receive either: 1) the positive affect intervention; or 2) a attention-matched control condition. Follow-up data will be collected at 3, 6, 12, and 15 months post-randomization. This RCT will provide an opportunity to examine the efficacy of an integrative intervention designed to promote long-term reductions in HIV viral load as the primary outcome. Secondary outcomes that will be examined include: increases positive affect, reductions in stimulant use, improvements in T-helper (CD4+) count, unsuppressed viral load, and decreases HIV transmission risk behavior. Identifying an efficacious intervention approach to decrease HIV viral load among methamphetamine-using MSM would substantially support the goals of the National HIV/AIDS Strategy to reduce HIV incidence and mitigate HIV-related health disparities.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Documentation of HIV-positive serostatus
* Speak English
* Biological verification of recent methamphetamine use
* Completion of at least three contingency management (CM) visits
* Self reported anal sex with a man (MSM) in the past 12 months

Exclusion Criteria:

* Inability to provide informed consent, evidenced by cognitive impairment
* HIV negative serostatus

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2018-10-08 (Actual); Study Completion 2018-10-08 (Actual)

PRIMARY OUTCOMES:
HIV Viral Load | 15 Months
  Log10 HIV viral load change and log10 viral load at 15 months

SECONDARY OUTCOMES:
Unsuppressed HIV viral load | 15 Months
  Any unsuppressed viral load (>= 200 copies/mL) over the 15-month follow-up period.
T-helper Count | 15 Months
  Change in T-helper (CD4+) count
Methamphetamine and Cocaine Use (Stimulant Use) | 15 Months
  Changes in methamphetamine and cocaine use (assessed via self-report and urine toxicology screening) over the 15-month follow-up.
Psychological Adjustment | 15 Months
  Changes in positive affect, negative affect, and depressive symptoms over the 15-month follow-up.
Potentially Amplified Transmission (PAT) Risk Behavior | 15 Months
  Changes in self-reported HIV transmission risk behavior with an unsuppressed HIV viral load (>= 200 copies/mL) over the 15-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: William Woods, Ph.D., Principal Investigator — University of California, San Francisco; Adam W. Carrico, Ph.D., Principal Investigator — Miami University; Judith T. Moskowitz, Ph.D., MPH, Principal Investigator — Northwestern University
Locations (1):
- Alliance Health Project, San Francisco, California, United States

REFERENCES:
- [Derived] Foley J, Batchelder AW, Bernier L, Glynn T, Moskowitz J, Carrico A. Facets of mindfulness are associated with inflammation biomarkers in a sample of sexual minority men with HIV. Psychol Health Med. 2025 Feb;30(2):368-383. doi: 10.1080/13548506.2024.2407445. Epub 2024 Sep 24. PMID 39315986
- [Derived] Carrico AW, Gomicronmez W, Jain J, Shoptaw S, Discepola MV, Olem D, Lagana-Jackson J, Andrews R, Neilands TB, Dilworth SE, Evans JL, Woods WJ, Moskowitz JT. Randomized controlled trial of a positive affect intervention for methamphetamine users. Drug Alcohol Depend. 2018 Nov 1;192:8-15. doi: 10.1016/j.drugalcdep.2018.07.029. Epub 2018 Sep 5. PMID 30195243
- [Derived] Carrico AW, Jain J, Discepola MV, Olem D, Andrews R, Woods WJ, Neilands TB, Shoptaw S, Gomez W, Dilworth SE, Moskowitz JT. A community-engaged randomized controlled trial of an integrative intervention with HIV-positive, methamphetamine-using men who have sex with men. BMC Public Health. 2016 Jul 30;16:673. doi: 10.1186/s12889-016-3325-1. PMID 27476110